CLINICAL TRIAL: NCT00875927
Title: Breezy Candy Halitosis Study
Brief Title: Effects of Breezy Candy on Halitosis
Acronym: BCHS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Breezy Industries Ltd. (Industry)
Responsible Party: Maya Eshed, CEO, Breezy Industries Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCHS
Record Dates: First submitted 2009-03-10; First posted 2009-04-06 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Halitosis
Keywords: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 - control (Active Comparator): candy not including scraping microcapsules
  Interventions: Other: no scraping microcapsules
- 2 - Scraping (Active Comparator): candy including scraping TCP microcapsules
  Interventions: Other: scraping microcapsules containing inert TCP microcapsules
- 3 - Scraping plus Propolis (Active Comparator): candy including scraping Propolis microcapsules
  Interventions: Other: scraping microcapsules containing Propolis
- 4 - Scraping plus Zinc (Active Comparator): candy including scraping Zinc microcapsules
  Interventions: Other: scraping microcapsules containing and Zinc
- 5 - Scraping plus Propolis and Zinc (Active Comparator): candy including scraping Propolis and Zinc microcapsules
  Interventions: Other: scraping microcapsules containing Propolis and Zinc

INTERVENTIONS:
Other: no scraping microcapsules — 1, 4 grams isomalt candy containing no scraping microcapsules
  Arms: 1 - control
Other: scraping microcapsules containing inert TCP microcapsules — 1, 4 grams isomalt candy containing 2% inert TCP scraping microcapsules
  Arms: 2 - Scraping
Other: scraping microcapsules containing Propolis — 1, 4 grams, isomalt candy containing 2% Propolis scraping microcapsules
  Arms: 3 - Scraping plus Propolis
Other: scraping microcapsules containing and Zinc — 1, 4 grams, isomalt candy containing 2% Zinc scraping microcapsules
  Arms: 4 - Scraping plus Zinc
Other: scraping microcapsules containing Propolis and Zinc — 1, 4 grams, isomalt candy containing 2% Propolis and Zinc scraping microcapsules
  Arms: 5 - Scraping plus Propolis and Zinc

SUMMARY:
Users of Breezy candy will utilize the candy's abrasiveness to scrape tongue surface. The scraping action together with the release of compounds contained inside the abrasive microcapsules will result in significant reduction of oral halitosis.

ELIGIBILITY:
Inclusion Criteria:

* adult
* healthy
* male
* female
* bad breath

Exclusion Criteria:

* subject suffering from Diabetes
* subject suffering from renal disease
* pregnant women
* cigarette smokers
* any illness of oral cavity for the last 3 months
* subjects undergoing chemotherapy
* treatment by antibiotic
* treatment by anti-inflammatory

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Users of Breezy Candy will have fresher breath over Control | 150 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Barak, MD, Principal Investigator — Mouth and Jaw institute, Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel